CLINICAL TRIAL: NCT07249827
Title: A Randomized Comparison Between 0.67 mcg/kg, 1 mcg/kg, and 1.33 mcg/kg of Perineural Dexmedetomidine for Ultrasound-Guided Infraclavicular Block
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Julián Aliste, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2025-11084
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Analgesia; Pain, Acute; Upper Extremity Surgery; Nerve Block
Keywords: Analgesia; Acute pain; Brachial plexus; Brachial plexus block; Postoperative pain; Nerve block
MeSH Terms: conditions — Agnosia; Acute Pain; Pain, Postoperative | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: blinded-randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A research assistant (licensed anesthesiologist) will prepare the local anesthetic solutions and will add the study drug following the randomization order. The operator, patient and investigator assessing the block will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 0.67 mcg/kg (Experimental): Addition of dexmedetomidine 0.67 mcg/kg to local anesthetics in infraclavicular brachial plexus block
  Interventions: Drug: dexmedetomidine (perineural) 0.67 mcg/kg
- 1 mcg/kg (Experimental): Addition of dexmedetomidine 1 mcg/kg to local anesthetics in infraclavicular brachial plexus block
  Interventions: Drug: dexmedetomidine (perineural) 1 mcg/kg
- 1.33 mcg/kg (Experimental): Addition of dexmedetomidine 1.33 mcg/kg to local anesthetics in infraclavicular brachial plexus block
  Interventions: Drug: dexmedetomidine (perineural) 1.33 mcg/kg

INTERVENTIONS:
Drug: dexmedetomidine (perineural) 0.67 mcg/kg — Perineural dexmedetomidine 0.67 mcg/kg will be added to the local anesthetic used to block the cords of the brachial plexus with an infraclavicular approach.
  Arms: 0.67 mcg/kg
Drug: dexmedetomidine (perineural) 1 mcg/kg — Perineural dexmedetomidine 1 mcg/kg will be added to the local anesthetic used to block the cords of the brachial plexus with an infraclavicular approach.
  Arms: 1 mcg/kg
Drug: dexmedetomidine (perineural) 1.33 mcg/kg — Perineural dexmedetomidine 1.33 mcg/kg will be added to the local anesthetic used to block the cords of the brachial plexus with an infraclavicular approach.
  Arms: 1.33 mcg/kg

SUMMARY:
This study will compare three different doses of perineural dexmedetomidine 0.67 mcg/kg, 1 mcg/kg, and 1.33 mcg/kg as adjuvants to local anesthetics for ultrasound-guided infraclavicular brachial plexus blocks (ICBs). Our research hypothesis is that 1.33 mcg/kg will provide a 15%-longer duration than 1mcg/kg, which in turn will provide a 15%-longer duration than 0.67 mcg/kg. Since analgesic duration and sensory duration can be influenced by intake of pain medications and surgical trauma to small cutaneous nerves, respectively, we will select motor block duration as the main outcome to better target the action of dexmedetomidine on the brachial plexus.

DETAILED DESCRIPTION:
With the approval of Ethics Committee of the McGill University Health Centre, a total of 69 patients undergoing upper extremity surgery (elbow and below) will be recruited. Recruitment will be carried out by an investigator not involved in patient care one day before surgery

All ICBs will be supervised by the coauthors and conducted preoperatively in an induction room.

After skin disinfection and draping, the ICB will be performed with a previously described technique. In each group, a proven 90% effective volume of 35 mL of local anesthetic solution will be injected. As LA solution, it will be used a mixture of lidocaine 1.0%-bupivacaine 0.25% with epinephrine 5 µ/mL plus PN 2 mg dexamethasone. The injectate will be slowly injected through the block needle.

Patients will be randomized to receive the study drug, PN dexmedetomidine 0.67 mcg/kg or PN dexmedetomidine 1 mcg/kg, or PN dexmedetomidine 1.33 mcg/kg mixed with the above-mentioned LA solution.

A research assistant (licensed anesthesiologist) will prepare the local anesthetic solutions and will add the study drug following the randomization order. The operator, patient, and investigator assessing the block will be blinded to group allocation.

The primary outcome will be the duration of the motor block (defined as the temporal interval between the end of LA injection through the block needle and the return of movement to the hand and fingers) for patients with successful ICBs. Patients will be provided with a data sheet and asked to record the time at which motor function returns. An investigator blinded to group allocation will collect this data sheet in person (inpatients) or by phone (outpatients) on postoperative day 1.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing upper limb surgery at or below the elbow
* age between 18 and 75 years
* American Society of Anesthesiologists classification 1-3
* body mass index between 18 and 35 kg/m2

Exclusion Criteria:

* adults who are unable to give their own consent
* allergy or contraindication to dexmedetomidine
* exposure to dexmedetomidine during the previous 48 hrs
* pre-existing neuropathy (assessed by history and physical examination)
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood workup i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or partial prothrombin time ≥ 50)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work-up i.e. creatinine. eGFR < 90)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work-up i.e. transaminases ≥ 100)
* allergy to LA
* pregnancy (as institutional policy, female patients with childbearing potential undergoing non urgent surgery are tested preoperatively for pregnancy with blood tests)
* breast feeding
* prior surgery in the infraclavicular region
* chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-12-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Motor block duration | 24-48 hours after block
  The elapsed period in minutes between the ending time of the local anesthetic injection and the time of return of hand and fingers movement

SECONDARY OUTCOMES:
Sensory block duration | 24-48 hours after block
  The elapsed period in minutes between the ending time of the local anesthetic injection and the time of the return of hand and fingers sensation
Analgesic block duration | 24-48 hours after block
  The elapsed period in minutes between the ending time of the local anesthetic injection and the time of the first sensation of pain in the surgical area
Block performance time | 1 hour before surgery
  Sum of: 1- the acquisition time of the ultrasonographic image. and 2- the time to perform the block itself (from the skin anesthesia to the end of local anesthetic injection)
Intensity of pain during block procedure | 1 hour before surgery
  Evaluated with the Numeric Rating Scale for Pain. This scale is graduated from 0 to 10 points. A 0-point score represents the absence of pain, and a 10-points score represents the worst imaginable pain. Patients will be asked to rate their pain verbally with this scale. The blinded assessor will register the score reported.
Block onset time | 1 hour before surgery
  Time required to reach a minimal sensorimotor composite score of 14 points out of a maximum of 16 points. The sensorimotor score is described in outcome 7.
Sensory and motor block score | 30 minutes after the ending time of local anesthetic injection
  The sensorimotor block will be assessed every 5 minutes until 30 minutes after the end of local anesthetic injection using a 16-point composite score evaluating sensory and motor block of musculocutaneous, medium, radial, and ulnar nerves.
  Sensation will be assessed with ice in each nerve territory with a 0 to 2 point scale. 0= no block, patients can feel cold; 1= analgesic block, the patient can feel touch but not cold; 2= anesthetic block, the patient cannot feel cold or touch.
  The motor function will be assessed for each nerve with a 0 to 2 points scale where 0= no motor block; 1= paresis; 2= paralysis.
  Successful blocks at 30 minutes correlate with a final score ( sum of all individual sensory and motor scores) of at least 14 points out of 16.
Incidence of complete block | 30 minutes after the ending time of local anesthetic injection
  Percentage of blocks with a minimal sensorimotor composite score of 14 points out of a maximum of 16 points at 30 minutes after the injection
Incidence of surgical anesthesia | 30-60 minutes after the ending time of local anesthetic injection
  Ability to proceed with surgery without the need for intravenous narcotics, general anesthesia, rescue blocks or local anesthesia infiltration by the surgeon
Incidence of nerve block side effects | 0 minutes after skin disinfection to 30 minutes after the nerve block
  Determined by the presence of paresthesia, local anesthetic systemic toxicity, vascular puncture, Horner syndrome, hoarseness, or pneumothorax after the block.
Respiratory depression | 30 minutes after the nerve block to 2 hours after surgery
  Presence of low respiratory rates (lower than 8 breaths per minute) or persistent oxygen requirements (pulse oximetry lower than 90% without supplementary oxygen).
  The respiratory rate and pulse oximetry are continuously measured intra- and post-operatively (in the post-anesthetic care unit) as a standard of care with a multiparameter monitor. Alarms are set to alert when predetermined levels are reached
Bradycardia | 30 minutes after the nerve block to 2 hours after surgery
  Defined as a heart rate lower than 50 beats per minute. The heart rate is continuously measured intra- and post-operatively (in the post-anesthetic care unit) as a standard of care with a multiparameter monitor. Alarms are set to alert when predetermined levels are reached
Hypotension | 30 minutes after the nerve block to 2 hours after surgery
  Mean arterial pressure lower than 60 mmHg. The blood pressure is measured intra- and post-operatively (in the post-anesthetic care unit) as a standard of care with a multiparameter monitor. Alarms are set to alert when predetermined levels are reached
Postoperative persistent sedation | 2 hours after surgery
  Persistent sedation after surgery using Ramsay sedation scale. The scale has 6 points from 1 to 6. A higher score represents a more sedated patient.
  1= anxious, agitated or restless; 2= co-operative, oriented and tranquil; 3= responds to command only; 4= brisk response to light pain or loud auditory stimulus; 5= sluggish response to light pain or loud auditory stimulus; 6= no response.
Persistent neurologic deficit | 7 days after surgery
  Presence of persistent sensory or motor postoperative deficit. The patients will be contacted by telephone and inquired about any sensory or motor deficit in the operated extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Julián Aliste, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo Y, Wang J, Jiang P, Wang D, Fan W, Yang X. Effect of erector spinae plane block with different doses of dexmedetomidine as adjuvant for ropivacaine on the postoperative quality of recovery after video-assisted thoracoscopic lobectomy surgery: a randomized controlled trial. BMC Anesthesiol. 2023 Aug 7;23(1):264. doi: 10.1186/s12871-023-02231-9. PMID 37550610
- [Background] Jung HS, Seo KH, Kang JH, Jeong JY, Kim YS, Han NR. Optimal dose of perineural dexmedetomidine for interscalene brachial plexus block to control postoperative pain in patients undergoing arthroscopic shoulder surgery: A prospective, double-blind, randomized controlled study. Medicine (Baltimore). 2018 Apr;97(16):e0440. doi: 10.1097/MD.0000000000010440. PMID 29668608
- [Background] Tran DQ, Dugani S, Dyachenko A, Correa JA, Finlayson RJ. Minimum effective volume of lidocaine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):190-4. doi: 10.1097/AAP.0b013e31820d4266. PMID 21270721
- [Background] Ouchi K. Dexmedetomidine 2 ppm Is Appropriate for the Enhancement Effect of Local Anesthetic Action of Lidocaine in Inferior Alveolar Nerve Block: A Preliminary, Randomized Cross-over Study. Clin J Pain. 2020 Aug;36(8):618-625. doi: 10.1097/AJP.0000000000000839. PMID 32398441
- [Background] Andersen JH, Jaeger P, Grevstad U, Estrup S, Geisler A, Vilhelmsen F, Dahl JB, Laier GH, Ilfeld BM, Mathiesen O. Systemic dexmedetomidine is not as efficient as perineural dexmedetomidine in prolonging an ulnar nerve block. Reg Anesth Pain Med. 2019 Mar;44(3):333-340. doi: 10.1136/rapm-2018-100089. Epub 2019 Jan 23. PMID 30679332
- [Background] Ouchi K, Sugiyama K. Dexmedetomidine Dose Dependently Enhances the Local Anesthetic Action of Lidocaine in Inferior Alveolar Nerve Block: A Randomized Double-Blind Study. Reg Anesth Pain Med. 2016 May-Jun;41(3):348-55. doi: 10.1097/AAP.0000000000000380. PMID 27015544
- [Background] Keplinger M, Marhofer P, Kettner SC, Marhofer D, Kimberger O, Zeitlinger M. A pharmacodynamic evaluation of dexmedetomidine as an additive drug to ropivacaine for peripheral nerve blockade: A randomised, triple-blind, controlled study in volunteers. Eur J Anaesthesiol. 2015 Nov;32(11):790-6. doi: 10.1097/EJA.0000000000000246. PMID 25695189
- [Background] Marhofer D, Kettner SC, Marhofer P, Pils S, Weber M, Zeitlinger M. Dexmedetomidine as an adjuvant to ropivacaine prolongs peripheral nerve block: a volunteer study. Br J Anaesth. 2013 Mar;110(3):438-42. doi: 10.1093/bja/aes400. Epub 2012 Nov 15. PMID 23161360
- [Background] Rancourt MP, Albert NT, Cote M, Letourneau DR, Bernard PM. Posterior tibial nerve sensory blockade duration prolonged by adding dexmedetomidine to ropivacaine. Anesth Analg. 2012 Oct;115(4):958-62. doi: 10.1213/ANE.0b013e318265bab7. Epub 2012 Jul 23. PMID 22826530
- [Background] Kim BS, Choi JH, Baek SH, Lee DH. Effects of Intraneural Injection of Dexmedetomidine in Combination With Ropivacaine in Rat Sciatic Nerve Block. Reg Anesth Pain Med. 2018 May;43(4):378-384. doi: 10.1097/AAP.0000000000000745. PMID 29505435
- [Background] Andersen JH, Grevstad U, Siegel H, Dahl JB, Mathiesen O, Jaeger P. Does Dexmedetomidine Have a Perineural Mechanism of Action When Used as an Adjuvant to Ropivacaine?: A Paired, Blinded, Randomized Trial in Healthy Volunteers. Anesthesiology. 2017 Jan;126(1):66-73. doi: 10.1097/ALN.0000000000001429. PMID 27792047
- [Background] Memari E, Hosseinian MA, Mirkheshti A, Arhami-Dolatabadi A, Mirabotalebi M, Khandaghy M, Daneshbod Y, Alizadeh L, Shirian S. Comparison of histopathological effects of perineural administration of bupivacaine and bupivacaine-dexmedetomidine in rat sciatic nerve. Exp Toxicol Pathol. 2016 Nov;68(10):559-564. doi: 10.1016/j.etp.2016.09.001. Epub 2016 Sep 17. PMID 27650364
- [Background] Brummett CM, Hong EK, Janda AM, Amodeo FS, Lydic R. Perineural dexmedetomidine added to ropivacaine for sciatic nerve block in rats prolongs the duration of analgesia by blocking the hyperpolarization-activated cation current. Anesthesiology. 2011 Oct;115(4):836-43. doi: 10.1097/ALN.0b013e318221fcc9. PMID 21666435
- [Background] Brummett CM, Amodeo FS, Janda AM, Padda AK, Lydic R. Perineural dexmedetomidine provides an increased duration of analgesia to a thermal stimulus when compared with a systemic control in a rat sciatic nerve block. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):427-31. doi: 10.1097/AAP.0b013e3181ef4cf0. PMID 20814283
- [Background] Brummett CM, Padda AK, Amodeo FS, Welch KB, Lydic R. Perineural dexmedetomidine added to ropivacaine causes a dose-dependent increase in the duration of thermal antinociception in sciatic nerve block in rat. Anesthesiology. 2009 Nov;111(5):1111-9. doi: 10.1097/ALN.0b013e3181bbcc26. PMID 19858875
- [Background] Brummett CM, Norat MA, Palmisano JM, Lydic R. Perineural administration of dexmedetomidine in combination with bupivacaine enhances sensory and motor blockade in sciatic nerve block without inducing neurotoxicity in rat. Anesthesiology. 2008 Sep;109(3):502-11. doi: 10.1097/ALN.0b013e318182c26b. PMID 18719449
- [Background] Tezuka M, Kitajima T, Yamaguchi S, Kimura Y, Hamaguchi S. Addition of dexmedetomidine prolongs duration of vasodilation induced by sympathetic block with mepivacaine in dogs. Reg Anesth Pain Med. 2004 Jul-Aug;29(4):323-7. doi: 10.1016/j.rapm.2004.03.004. PMID 15305251
- [Background] Poree LR, Guo TZ, Kingery WS, Maze M. The analgesic potency of dexmedetomidine is enhanced after nerve injury: a possible role for peripheral alpha2-adrenoceptors. Anesth Analg. 1998 Oct;87(4):941-8. doi: 10.1097/00000539-199810000-00037. PMID 9768799
- [Background] Abdulatif M, Fawzy M, Nassar H, Hasanin A, Ollaek M, Mohamed H. The effects of perineural dexmedetomidine on the pharmacodynamic profile of femoral nerve block: a dose-finding randomised, controlled, double-blind study. Anaesthesia. 2016 Oct;71(10):1177-85. doi: 10.1111/anae.13603. PMID 27611039
- [Background] Ghazaly HF, Aly AAA, Zaher ZZ, Hassan MM, Mahmoud AA. Comparison of the efficacy of two doses of dexmedetomidine as an adjunct to levobupivacaine in infraclavicular brachial plexus block: prospective double-blinded randomized controlled trial. BMC Anesthesiol. 2022 Nov 5;22(1):338. doi: 10.1186/s12871-022-01858-4. PMID 36335297
- [Background] Bravo D, Aliste J, Layera S, Fernandez D, Leurcharusmee P, Samerchua A, Tangjitbampenbun A, Watanitanon A, Arnuntasupakul V, Tunprasit C, Gordon A, Finlayson RJ, Tran DQ. A multicenter, randomized comparison between 2, 5, and 8 mg of perineural dexamethasone for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2019 Jan;44(1):46-51. doi: 10.1136/rapm-2018-000032. PMID 30640652
- [Background] Aliste J, Layera S, Bravo D, Aguilera G, Erpel H, Garcia A, Lizama M, Finlayson RJ, Tran D. Randomized comparison between perineural dexamethasone and combined perineural dexamethasone-dexmedetomidine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2022 Jun 21:rapm-2022-103760. doi: 10.1136/rapm-2022-103760. Online ahead of print. PMID 35728840
- [Background] Aliste J, Layera S, Bravo D, Fernandez D, Jara A, Garcia A, Finlayson RJ, Tran DQ. Randomized comparison between perineural dexamethasone and dexmedetomidine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2019 Jul 11:rapm-2019-100680. doi: 10.1136/rapm-2019-100680. Online ahead of print. PMID 31300595